CLINICAL TRIAL: NCT06015412
Title: Effects Of Osteoarthritis Grades On Pain, Function, And Quality Of Life
Brief Title: Physical Parameters in Osteoarthritis Stages
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Emine Cihan, Asst. Prof, Selcuk University
Other Study IDs: 2023/11-21
Record Dates: First submitted 2023-08-21; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis; Pain; Quality of Life
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Grade 1 osteoarthritis: disease stages 1 according to the Kellgren-Lawrence radiographic classification system
  Interventions: Diagnostic Test: Radiographic classification
- Grade 2 osteoarthritis: disease stages 2 according to the Kellgren-Lawrence radiographic classification system
  Interventions: Diagnostic Test: Radiographic classification
- Grade 3 osteoarthritis: disease stages 3 according to the Kellgren-Lawrence radiographic classification system
  Interventions: Diagnostic Test: Radiographic classification
- Grade 4 osteoarthritis: disease stages 4 according to the Kellgren-Lawrence radiographic classification system
  Interventions: Diagnostic Test: Radiographic classification

INTERVENTIONS:
Diagnostic Test: Radiographic classification — disease stages ranged from 1 to 4 according to the Kellgren-Lawrence radiographic classification system

SUMMARY:
To investigate the extent to which pain, functionality, and quality of life change over the progression of osteoarthritis grades.

ELIGIBILITY:
Inclusion Criteria:

* having the same OA grade in both knees
* volunteering to participate in the study
* not having undergone previous lower extremity surgery

Exclusion Criteria:

* neurological disorders;
* those with a history of surgery related to the lower extremities;
* those with orthopedic problems in the lower extremities, such as tendinopathy and bursitis;
* those who had neurological, orthopedic, or cognitive disorders that would prevent walking;
* those with a diagnosis of diabetes, obesity, or rheumatological disorders;
* those who had received intra-articular injection therapy within the last three months;
* and those with malignancy or perception problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diagnosed with the same grade of knee OA in both knees by the responsible physician in the hospital
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 2 minutes
  a 10-cm straight line with 0 on one end indicating no pain and 10 on the other end signifying unbearable pain. The participants were asked to mark the intensity of their current pain on the line
two-minute walk test (2MWT) | 2 minutes
  A 45-meter corridor was used for the 2MWT. The start and end points were marked, and the participants were asked to walk at a normal pace within these boundaries. The distance covered in two minutes was recorded
Western Ontario and McMaster Universities Osteoarthritis Index | 10 minutes
  The questionnaire consists of 24 items, each scored from 0 to 4. The total score is obtained by summing the point equivalents of the responses given to all items. A higher score indicates poorer functionality
Nottingham Health Profile (NHP) | 10 minutes
  This tool comprises 38 questions in six domains, namely energy, pain, social isolation, physical mobility, emotional reactions, and sleep. Each domain is scored from 0 to 100. The total score is obtained by summing the scores obtained from the six domains. High scores indicate a good quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No